CLINICAL TRIAL: NCT05628480
Title: Multi-omics Analyses Reveal Microbiota-gut-brain Axis in ICU Patients With Post-cardiac Surgery Delirium
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: National Clinical Research Center for Cardiovascular Diseases, Fuwai Hospital, Chinese Academy of Medical Sciences (Unknown)
Responsible Party: Sponsor
Other Study IDs: NCRC2010010
Record Dates: First submitted 2022-11-07; First posted 2022-11-28 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Delirium; Cardiac Disease; Gastrointestinal Microbiome
MeSH Terms: conditions — Emergence Delirium; Heart Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POD group: According to RASS and CAM-ICU scales, patients who suffer from post-cardiac surgery delirium in ICU will be include into POD group
- Non-POD group: According to RASS and CAM-ICU scales，patients who do not judge as post-cardiac surgery delirium in ICU will be include into non-POD group

SUMMARY:
This case-control study is planned to recruit patients who meet the enrollment conditions, receive cardiac surgery (cardiac valve surgery or coronary artery bypass surgery) and cardiopulmonary bypass, and sign the informed consent form in the second ward of adult cardiac surgery, Fuwai Hospital. Use RASS, CAM-ICU scales to evaluate postoperative patients and divide them into delirium and non-delirium groups according to whether they had delirium after surgery. There will be 30 patients in each group. Match the two groups in terms of surgical type, duration of cardiopulmonary bypass, gender and age range (± 3 years). Collect and record the preoperative, intraoperative and postoperative data of the enrolled patients, including cardiopulmonary bypass time, ICU stay time, length of mechanical ventilation, hemodynamics and other data. Fecal and/or blood samples are collected from 60 patients before, immediately after and after operation.

The laboratory test and analysis shall be started after the collection of clinical samples. Fecal samples are used for Metagenomics Sequencing and Functional genomics. Blood samples are analyzed by serum metabolomics for changes in intestinal metabolites entering the blood circulation. Simultaneous measurement of IL-6 and TNF in peripheral blood with serum samples- α, IL-1a,IFN-γ and LPS, D-lactic acid and diamine oxidase levels.Use Multi-omics approach to analyze the correlation between intestinal flora diversity, functional gene abundance and blood metabolites, inflammation level and intestinal barrier function, and to find the clinical evidence of the correlation between microbiota-gut-brain axis and the occurrence of POD in patients. Through comprehensive analysis of the research results of this experiment, access to literature, write papers, submit papers and publish relevant papers.

ELIGIBILITY:
Inclusion Criteria:

* elective cardiac valve surgery or coronary artery bypass grafting
* open heart surgery under hypothermic cardiopulmonary bypass under intravenous and/or inhalation general anesthesia
* No history of delirium attack, no cognitive impairment, normal speech, and certain ability of speaking and reading
* age>18
* Informed consent of patients, voluntary participation (or consent of family members), and signing of informed consent

Exclusion Criteria:

* There are organic brain diseases (preoperative brain CT examination)
* Hearing or visual impairment that may affect delirium assessment
* Suspected or confirmed history of alcohol/drug/drug abuse
* Previous history of mental illness or preoperative use of antipsychotic drugs
* Moderate and severe renal function damage (blood creatinine > 2mg/dL or 177mmol/L) or abnormal liver function (alanine aminotransferase>2 times the upper limit of normal value) or other serious lung diseases
* Hematologic diseases, bone marrow and/or lymphoid diseases, leukopenia
* Use immunosuppressive drugs or autoimmune diseases
* Pregnant
* Accompanied by other diseases that may affect their survival, such as tumor
* HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who meet the enrollment conditions, receive cardiac surgery (heart valve surgery or coronary artery bypass surgery) and cardiopulmonary bypass (CPB) in the Department of Cardiovascular Surgery, Fuwai Hospital, Chinese Academy of Medical Sciences.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
postoperative delirium | 1-4 days after cardiac surgery
  Use the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) to identify delirium in critically ill patients.The CAM-ICU consists of four main components:inattention, autonomic instability, disorganized thinking, altered level of consciousness.If patient have 1) acute onset of mental status changes or a fluctuating course and 2)inattention and 3)disorganized thinking or 4)altered level of consciousness, thus the patient can be assessed as postoperative delirium (1+2+3/4=POD).
type of postoperative delirium | 1-4 days after cardiac surgery
  The Richmond Agitation Sedation Scale (RASS) is an instrument designed to assess the level of alertness and agitated behavior in critically-ill patients.The RASS is a 10-point scale ranging from -5 to +4. Levels -1 to -5 denote 5 levels of sedation, levels +1 to +4 describe increasing levels of agitation,level 0 is "alert and calm." 1.Hyperactive POD: postoperative delirium patient with RASS scores +1~+4; 2.Hypoactive POD:Hyperactive POD: postoperative delirium patient with RASS scores -3~0; 3.Mixed POD: postoperative delirium patient with RASS score fluctuate between positive and negative.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided